CLINICAL TRIAL: NCT01441232
Title: A Phase 1, Open-label, 3-period, 3-treatment, Single Dose Crossover Study to Evaluate the Pharmacodynamic Effects of LX4211 When Administered Concurrently With JANUVIA® (Sitagliptin) in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Pharmacodynamic Effects of Single-Dose Co-Administration of LX4211 With Januvia® in Type 2 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LX4211.1-105-DM; LX4211.105 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental)
  Interventions: Drug: LX4211
- Treatment C (Experimental)
  Interventions: Drug: LX4211; Drug: Januvia®
- Treatment B (Active Comparator)
  Interventions: Drug: Januvia®

INTERVENTIONS:
Drug: LX4211 — 400 mg of LX4211 administered as two 200 mg tablets
  Arms: Treatment A; Treatment C
Drug: Januvia® — 100 mg Januvia® (sitagliptin) administered as one 100 mg sitagliptin tablet
  Arms: Treatment B; Treatment C

SUMMARY:
This study is intended to evaluate the pharmacodynamics, safety, and tolerability of LX4211 when administered concurrently with sitagliptin (Januvia®) in patients with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years of age
* History of Type 2 Diabetes Mellitus for at least 3 months prior to Screening, with HgbA1c values of 6.5 to 10.5% and C-peptide ≥1.0 ng/mL
* Body mass index (BMI) ≤45 kg/sq m
* Willing and able to self-monitor blood glucose
* Able to provide written informed consent

Exclusion Criteria:

* History of Type 1 diabetes mellitus, diabetic ketoacidosis, hyperosmolar nonketotic syndrome, or diabetes resulting from pancreatic disorder or secondary diabetes
* Current use of any blood glucose lowering agent other than metformin
* History of renal disease or clinically significant abnormal kidney function tests at Screening or Day -2
* Presence of active hepatic disease or clinically significant abnormal liver function tests at Screening or Day -2
* History of myocardial infarction, severe/unstable angina, or coronary revascularization procedure within 6 months of Day -2
* History of clinically significant cardiac arrhythmias within 1 year of Day -2
* Congestive heart failure and/or New York Heart Association (NYHA) class III or IV symptoms of heart failure
* Subjects with uncontrolled Stage 3 hypertension
* History of 2 or more emergency room visits, doctor's visits, or hospitalizations due to hypoglycemia within 6 months of Day -2
* History of alcohol or drug abuse within 12 months of Screening
* History of bowel resection > 20 cm, any malabsorptive disorder, severe gastroparesis, and GI procedure for the purpose of weight loss that would slow gastric emptying
* History of HIV or hepatitis C
* Major surgery within 3 months of Day -2 or any planned surgery during the study
* History of any active infection within 2 weeks of Day -2
* History of pancreatitis
* History of any malignancy within the last 5 years which would affect the diagnosis or assessment of LX4211 or sitagliptin
* History of any serious adverse reaction or hypersensitivity to LX4211 or sitagliptin
* Presence of any clinically significant physical, laboratory, or ECG findings or any concurrent condition at Screening that may interfere with the study in the opinion of the investigator
* Triglycerides > 1000 mg/dL at Screening or Day -2
* Donation or loss of >400 mL of blood or blood product within 8 weeks prior to Day -2
* Use of any tobacco product for the duration of study participation
* Use of corticosteroids within 2 weeks of Day 1
* Use of digoxin or warfarin within 2 weeks prior to Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in gut hormones | Days 1, 8, and 15

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose | Days 1, 8, and 15
Change from baseline in postprandial glucose | Days 1, 8, and 15
Change from baseline in insulin | Days 1, 8, and 15
Change from baseline in peptide YY | Days 1, 8, and 15
Change from baseline in urinary glucose excretion | Days 1, 8, and 15

CONTACTS AND LOCATIONS:
Overall Officials: Ikenna Ogbaa, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, San Antonio, Texas, United States

REFERENCES:
- [Derived] Zambrowicz B, Ding ZM, Ogbaa I, Frazier K, Banks P, Turnage A, Freiman J, Smith M, Ruff D, Sands A, Powell D. Effects of LX4211, a dual SGLT1/SGLT2 inhibitor, plus sitagliptin on postprandial active GLP-1 and glycemic control in type 2 diabetes. Clin Ther. 2013 Mar;35(3):273-285.e7. doi: 10.1016/j.clinthera.2013.01.010. Epub 2013 Feb 21. PMID 23433601